CLINICAL TRIAL: NCT06626906
Title: Predictive Value of Sleep Apnea-specific Pulse Transit Time Response for Incident Subclinical Abnormalities in Left Ventricle Structure and Function in Cohort of moderate-to Severe Obstructive Sleep Apnea
Brief Title: Predictive Value of Sleep Apnea-specific PTT Response for Incident Subclinical Abnormalities in LV Structure and Function in Cohort of moderate-to Severe OSA
Status: Completed | Type: Observational
Sponsor: Xu J (Other)
Collaborators: The first affiliated Hospital of Nanjing Medical University, Jiangsu Province (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Xu J, Chief physician, Associate professor, Huai'an No.1 People's Hospital
Organization: Huai'an No.1 People's Hospital (Other)
Other Study IDs: YX-Z-2023-027-01
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: retrospective cohort; multicenter studies; observational study model
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography, Blood sampling for biomarker assays

SUMMARY:
This observational study aims to provide evidence for identifying those who mostly suffer from LV injury and will help construct an optimal strategy for clinical practice. The main question it aims to answer is:

Could acute PTT response surrounding obstructive respiratory events predict the incidence of subclinical abnormalities in LV structure and function in moderate-to-severe OSA patients? Participants who had undergone standard polysomnography and were diagnosed with moderate-to-severe OSA 5 years ago were required to complete the cardiac remodeling and function evaluation.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a widely prevalent medical condition characterized by recurrent upper airway obstruction with intermittent hypoxia, sleep disruption, and increased ventilation. Serial studies have shown that OSA promotes oxidative stress, sympathetic activity, and intrathoracic pressure fluctuation, resulting in adverse cardiac structures and function. The cumulative data from observational studies have linked the apnea-hypopnea index (AHI), an indicator of OSA severity, with increased LV injury. As OSA is a highly heterogeneous disorder, with diverse pathways to disease, expression of disease, susceptibility to co-morbidities, and response to therapy. Hence, OSA is ideally suited to precision medicine approaches. While the current assessment relies on the AHI, this traditional metric poorly reflects the complex pathophysiological of OSA on cardiac injury.

Asymptotic cardiac dysfunction is not easily identified, and many sufferers remain undiagnosed in clinical practice. Focusing on recognition and treatment of subclinical cardiac injury early is a potentially powerful strategy to prevent progression to clinical or symptomatic heart failure. In OSA patients, the BP and heart rate (HR) changes occurring with obstructive events involve an initial decrease early in the event, a gradual increase during the terminal portion of the event, and an immediate surgeon resumption of ventilation. These acute hemodynamic and autonomic changes may be closely associated with the development and progression of cardiovascular disease. Whether this OSA-specific cardiovascular reactivity pattern is the potentially early warning indicator of cardiac injury is unknown.

A physiologic parameter termed pulse transit time (PTT) has been studied intensively as an indirect marker for variations in cardiovascular-related reactivity. It can be generally referred to as the time difference for a pulse wave to travel between two arterial sites. The speed at which this arterial pressure wave travels was used to assess nocturnal blood pressure variation, arterial stiffness changes, autonomic nervous response, and inspiratory effort. More experimentally focused investigations with PTT as a key measure in cardiovascular-related studies are being reported.

In the present study, the investigators examined acute PTT changes surrounding obstructive events, for PTT can be easily measured in standard polysomnography (PSG). The investigators hypothesized that the specific respiratory events PTT response would predict incident subclinical abnormalities in LV structure and function in a cohort of moderate-to-severe OSA without other confounded morbidities. The results of this study provide evidence for identifying those who mostly suffer from LV injury and will help construct an optimal strategy for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Moderate to severe OSA(AHI≥15 times/hour).

Exclusion Criteria:

1. baseline hypoxia;
2. other sleep disorders;
3. received regular CPAP treatment(on average of ≥ 4 hours for CPAP use per night during the retrospective period);
4. the prevalent diseases at baseline might have influenced the results of echocardiographic results: hypertension chronic atrial fibrillation, atrioventricular block, bundle branch blocks, a permanent pacemaker, heart failure, valvular heart disease, pulmonary emboli, abnormal thyroid function, cardiomyopathies, pulmonary hypertension, use of digitalis, use of antiarrhythmic agents, use of beta-blockers, or use of calcium agonists affecting heart rate (HR), including verapamil and diltiazem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients aged 18 years and older, with moderate-to-severe OSA, who were diagnosed between January 1 2014, and December 31 2019 at The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, the First Affiliated Hospital of Nanjing Medical University, and the Affiliated Hospital of Xuzhou Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
the cardiac remodeling evaluation | from October 2023 to May 2024
  The echocardiogram was carried out using machines equipped with a 2.5-MHz probe. All 2D and Doppler images and measurements were obtained in agreement with the European Association of Echocardiography/American Society of Echocardiography guidelines.
  Measures of LV remodeling included LV end-systolic (LVDs) in centimeters, and end-diastolic diameter (LVDd) in centimeters, interventricular septum thickness at end-diastole (IVSd) in centimeters, LV mass (LVM) in grams. LVM (LVMI) was calculated as the ratio of LVM in grams and body surface area in square meters. LVH was defined as an LVMI of 111 g/m2or 50 g/m2 in males and of 106 g/m2or 47 g/m2 in females.
the cardiac function evaluation | from October 2023 to May 2024
  The echocardiogram was carried out using machines equipped with a 2.5-MHz probe. All 2D and Doppler images and measurements were obtained in agreement with the European Association of Echocardiography/American Society of Echocardiography guidelines.
  Measures of LV diastolic function included the average of the septal and lateral mitral annular descent tissue Doppler velocity (E') in cm/s, early mitral inflow velocity E' in cm/s, and the ratio of E/E'. Measures of systolic function included LV ejection fraction (EF) in percentage using Simpson biplane method of disks in 2-chamber and 4-chamber apical views (a single view was used in cases where one view was technically suboptimal).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drager LF, Bortolotto LA, Figueiredo AC, Silva BC, Krieger EM, Lorenzi-Filho G. Obstructive sleep apnea, hypertension, and their interaction on arterial stiffness and heart remodeling. Chest. 2007 May;131(5):1379-86. doi: 10.1378/chest.06-2703. PMID 17494787
- [Result] Alomri RMA, Kennedy GA, Wali S, Alhejaili F, Zelko M, Robinson SR. Association between cognitive dysfunction and nocturnal peaks of blood pressure estimated from pulse transit time in obstructive sleep apnoea. Sleep Med. 2022 Feb;90:185-191. doi: 10.1016/j.sleep.2022.01.005. Epub 2022 Jan 10. PMID 35183866
- [Result] Nisbet LC, Yiallourou SR, Nixon GM, Biggs SN, Davey MJ, Trinder J, Walter LM, Horne RS. Characterization of the acute pulse transit time response to obstructive apneas and hypopneas in preschool children with sleep-disordered breathing. Sleep Med. 2013 Nov;14(11):1123-31. doi: 10.1016/j.sleep.2013.06.010. Epub 2013 Aug 3. PMID 24047534
- [Result] Nisbet LC, Nixon GM, Yiallourou SR, Biggs SN, Davey MJ, Trinder J, Walter LM, Horne RS. Sleep-disordered breathing does not affect nocturnal dipping, as assessed by pulse transit time, in preschool children: evidence for early intervention to prevent adverse cardiovascular effects? Sleep Med. 2014 Apr;15(4):464-71. doi: 10.1016/j.sleep.2013.11.787. Epub 2014 Feb 10. PMID 24684978
- [Result] Foo JY, Wilson SJ, Williams GR, Harris MA, Cooper DM. Pulse transit time changes observed with different limb positions. Physiol Meas. 2005 Dec;26(6):1093-102. doi: 10.1088/0967-3334/26/6/018. Epub 2005 Nov 7. PMID 16311456
- [Result] Kwon Y, Jacobs DR Jr, Lutsey PL, Brumback L, Chirinos JA, Mariani S, Redline S, Duprez DA. "Sleep disordered breathing and ECG R-wave to radial artery pulse delay, The Multi-Ethnic Study of Atherosclerosis". Sleep Med. 2018 Aug;48:172-179. doi: 10.1016/j.sleep.2018.05.005. Epub 2018 May 21. PMID 29960211
- [Result] Foo JY, Lim CS. Pulse transit time as an indirect marker for variations in cardiovascular related reactivity. Technol Health Care. 2006;14(2):97-108. PMID 16720953
- [Result] Parish JM, Somers VK. Obstructive sleep apnea and cardiovascular disease. Mayo Clin Proc. 2004 Aug;79(8):1036-46. doi: 10.4065/79.8.1036. PMID 15301332
- [Result] Imadojemu VA, Gleeson K, Gray KS, Sinoway LI, Leuenberger UA. Obstructive apnea during sleep is associated with peripheral vasoconstriction. Am J Respir Crit Care Med. 2002 Jan 1;165(1):61-6. doi: 10.1164/ajrccm.165.1.2009062. PMID 11779731
- [Result] Ogilvie RP, Genuardi MV, Magnani JW, Redline S, Daviglus ML, Shah N, Kansal M, Cai J, Ramos AR, Hurwitz BE, Ponce S, Patel SR, Rodriguez CJ. Association Between Sleep Disordered Breathing and Left Ventricular Function: A Cross-Sectional Analysis of the ECHO-SOL Ancillary Study. Circ Cardiovasc Imaging. 2020 May;13(5):e009074. doi: 10.1161/CIRCIMAGING.119.009074. Epub 2020 May 15. PMID 32408831
- [Result] Bradley TD, Floras JS. Sleep apnea and heart failure: Part I: obstructive sleep apnea. Circulation. 2003 Apr 1;107(12):1671-8. doi: 10.1161/01.CIR.0000061757.12581.15. No abstract available. PMID 12668504
- [Result] Gottlieb DJ, Yenokyan G, Newman AB, O'Connor GT, Punjabi NM, Quan SF, Redline S, Resnick HE, Tong EK, Diener-West M, Shahar E. Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study. Circulation. 2010 Jul 27;122(4):352-60. doi: 10.1161/CIRCULATIONAHA.109.901801. Epub 2010 Jul 12. PMID 20625114